CLINICAL TRIAL: NCT05535153
Title: Reproducibility of the Functional Movement Screen Test in the Normandy Amateur Rugby Player
Brief Title: Reproducibility of the Functional Movement Screen Test
Status: Completed | Type: Observational
Sponsor: Pole Sante Grace de Dieu (Other)
Responsible Party: Principal Investigator, Guillaume GALLIOU, Principal Investigator, Pole Sante Grace de Dieu
Other Study IDs: 20220101
Record Dates: First submitted 2022-08-16; First posted 2022-09-10 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Locomotor Pain Disorder
Keywords: FMS, rugby
MeSH Terms: conditions — Collagen Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experime: Hurdle steps Deep squats Inline lunges Shoulder Clearing Active straight leg raise Trunk stability pushup Rotary stability Spinal extension exam Spinal flexion exam
  Interventions: Other: functional movement screen

INTERVENTIONS:
Other: functional movement screen — The volunteer subjects had to perform the FMS test at the request of the investigator, which is made up of seven movements: the squat, the crossing of the hurdle, the line lunge, the active elevation with the straight leg, a movement concerning the mobility of the shoulders, a rotational stability assessment movement and a core stability assessment movement.

SUMMARY:
The main objective of the study is to determine the inter-evaluator and intra-evaluator reproducibility of the FMS test as an evaluation tool in amateur rugby players.

The secondary objective of the study is to evaluate the abilities of the FMS test as a predictive tool for detecting possible injuries during a sports season in amateur rugby players.

DETAILED DESCRIPTION:
Rugby is a very popular sport in France, since it has more than 300,000 dismissed. The 2023 World Cup will take place in France, and in view of the enthusiasm that is created around the "XV de France" team, there will be a great number of new players. Yet there are many injuries in this sport, despite the adaptations of the French Rugby Federation. The injuries of these amateur players will handicap their performance within their club (an injured player will be injured more easily in the future) and have a impact on their personal and professional life. With this in mind, it would be desirable to have a predictive tool for possible wounds. For this, Agullo et al. had in the previous study "Reproducibility of the Functional Movement Screen (FMS) test in the amateur Rugby player" (ID-RCB: 2018-A03490-55) selected this tool already evaluated in the context of prediction injuries in other sports (hockey or American football). The FMS offers an overall assessment of the subject, based on seven so-called movements fundamentals, combining mobility and stability, making it possible to assess the deficiencies of the individual; a prevention plan will then be adapted to the subject.

ELIGIBILITY:
Inclusion Criteria:

* Rugby players in the "Amateur" and "Senior" categories
* Must be able to play a match within a week of the FMS test evaluation.

Exclusion Criteria:

* players evolving or having evolved beyond the "Federal 3" division for men or "Federal 1" for women
* Pregnant and breastfeeding women
* People in an emergency situation
* People unable to give their consent (including people under guardianship)
* Patients already involved in another study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The subjects recruited are rugby players aged 18 to 55, playing or having played in the "Amateur" and "Senior" categories.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Functional Movement Screen | 1 year
  Intraclass correlation coefficient with data : FMS score between rater one and rater two

SECONDARY OUTCOMES:
Functional Movement Screen | through study completion, an average of 1 year
  Functional Movement Screen (FMS) will be used as a assessment tool to screen the risk of injury in rugby

CONTACTS AND LOCATIONS:
Locations (1):
- PSLA GDD, Caen, France

IPD SHARING:
Plan to Share IPD: No